CLINICAL TRIAL: NCT06269068
Title: Does Central Sensitization Mediate Neuropathic Complaints in Lumbar Disc Herniation? A Cross-sectional Observational Study
Brief Title: Investigation of the Relationship Between Central Sensitization and Neuropathic Pain in Lumbar Disc Herniation
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 12.01.2024.10
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Central Sensitisation
Keywords: Central sensitisation; Lumbar Disc Herniation; Neuropathic Pain; Central sensitization inventory
MeSH Terms: conditions — Intervertebral Disc Displacement; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with lumbar disc herniation
  Interventions: Diagnostic Test: Central sensitization inventory; Other: Short form-36; Other: Oswestry Low Back Pain Disability Questionnaire; Other: Douleur Neuropathique 4; Other: Visual analogue scale

INTERVENTIONS:
Diagnostic Test: Central sensitization inventory — Standardized questionnaire to determine the level of central sensitization. Patients with a score of 40 and above are considered to have central sensitization.
  Other Names: CSI
Other: Short form-36 — Standardized questionnaire to investigate the quality of life in patients. The score of the scale is between 0-100. The higher scores are associated with greater deterioration in quality of life.
  Other Names: SF-36
Other: Oswestry Low Back Pain Disability Questionnaire — With this scale, it is questioned to what extent the patient is affected by low back pain in selected daily living activities under certain ten headings. In total scoring, disability is expressed as a percentage, and high scores are interpreted in favor of an increase in disability.
  Other Names: ODI
Other: Douleur Neuropathique 4 — The questionnaire consists of 10 items; while the nature of pain is questioned in 7 items, the other 3 items include brief sensory examination. Patients with a score of 4 or more out of 10 are considered to have neuropathic pain.
  Other Names: DN4
Other: Visual analogue scale — global pain score on a 0 to 10
  Other Names: VAS

SUMMARY:
Central sensitization (CS) is as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with in many musculoskeletal diseases with chronic pain has been demonstrated in several studies. CS is also one of the main mechanisms proposed in the generation of neuropathic pain, and the relationship between pain sensitization and neuropathic complaints has been shown in different diseases.In this study, it was aimed to investigate the effect of central sensitization on the distribution pattern and neuropathic character of pain in patients with lumbar disc herniation who applied to the physical medicine and rehabilitation outpatient clinic.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is one of the leading causes of musculoskeletal pain and its lifetime prevalence is around 80%. Different types of pain can be seen in patients with LDH, which are classified by the International Association for the Study of Pain (IASP) as nociceptive low back pain, somatic referred pain, radicular pain, and radiculopathy. While nociceptive low back pain originates from the structures in the lumbar spine, this pain is characterized as somatic referred pain when it spreads to the lower extremities. Radicular pain is different from these two pains in mechanism and character, and neuropathic complaints accompany axial pain. LDH is also the most common cause of lumbar radicular pain and causes neuropathic pain by irritation of the spinal nerve or dorsal root ganglion. In recent studies, it has been shown that nociceptor hyperexcitability and continuous stimulus discharge into the central nervous system play an important role in the formation of neuropathic pain. This mechanism is also encountered in central sensitization (CS), which is well-known to be associated with chronic pain and characterized by increased response to painful stimuli. Although there are many definitions of CS in the literature, one of the most comprehensive definitions was made as "Changes in the membrane excitability of the central pain pathways and changes in the synaptic transmission of the dorsal anterior horn cells and a decrease in the inhibition of the descending pathways". In animal models, inflammation-mediated spinal microglia activation has been shown to play a role in chronic radicular pain secondary to disc herniation, which has been associated with the development of central sensitization. A study showed that the frequency of CS is increased in patients with chronic low back pain, and this rate is variable in patients with LDH. In addition, data on the role of CS in LDH-related pain, especially radicular pain, are increasing.Considering all these data, CS is likely to affect pain in various ways in patients with LDH, particularly in its severity, extent, and neuropathic component. Therefore, in this study, it was aimed to investigate the relationship between CS accompanying LDH patients with pain characteristics and neuropathic pain development.

ELIGIBILITY:
Inclusion Criteria:

Having a diagnosis of lumbar disc herniation Accepting to participate in the study

Exclusion Criteria:

Concomitant active systemic inflammatory disease, infection and malignancy Having disease that will cause neuropathic pain in the other lower extremity, such as polyneuropathy, multiple sclerosis etc Refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients aged 18-65 years diagnosed with lumbar disc herniation will be recruited from a PMR outpatient clinic of a state hospital
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | 6 months
  25 somatic and psychosocial symptoms, which are frequently found in patients with central sensitization in part A, are questioned. In part B, the presence of diseases whose relationship with central sensitization is well defined is questioned in the patient without participating in scoring. Central sensitization is assumed in patients who score 40 or more over 100 points.
DN4 | 6 months
  The DN4 scale was developed in 2005 to detect the neuropathic component of pain.This questionnaire consists of 10 items; While the nature of pain is questioned in 7 items, the other 3 items include brief sensory examination. Patients with a score of 4 or more out of 10 are considered to have neuropathic pain.

SECONDARY OUTCOMES:
VAS pain | 6 months
  The patients pain severity will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
SF-36 | 6 months
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health.The scale was developed by Ware in 1987 and consists of 36 questions questioning 8 sub-parameters regarding the health status of the person.These parameters are physical function, pain, limitation due to physical and emotional problems, emotional well-being, social function, fatigue and general health perception.
ODI | 6 months
  This scale was developed for assessing the severity of disability in chronic low back pain patients. This scale consists of 10 items that evaluates the limitation of daily life activities of patients in the last month.It is accepted that the higher the score, the higher disability.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Şanal Toprak, Asst.Prof, Study Chair — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Fevzi Çakmak Mah, Muhsin Yazıcıoğlu Cd, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author, upon reasonable request.

REFERENCES:
- [Background] Al Qaraghli MI, De Jesus O. Lumbar Disc Herniation. 2023 Aug 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560878/ PMID 32809713
- [Background] Bogduk N. On the definitions and physiology of back pain, referred pain, and radicular pain. Pain. 2009 Dec 15;147(1-3):17-9. doi: 10.1016/j.pain.2009.08.020. Epub 2009 Sep 16. No abstract available. PMID 19762151
- [Background] Dower A, Davies MA, Ghahreman A. Pathologic Basis of Lumbar Radicular Pain. World Neurosurg. 2019 Aug;128:114-121. doi: 10.1016/j.wneu.2019.04.147. Epub 2019 Apr 25. PMID 31028982
- [Background] Meacham K, Shepherd A, Mohapatra DP, Haroutounian S. Neuropathic Pain: Central vs. Peripheral Mechanisms. Curr Pain Headache Rep. 2017 Jun;21(6):28. doi: 10.1007/s11916-017-0629-5. PMID 28432601
- [Background] Huang Y, Li Y, Zhong X, Hu Y, Liu P, Zhao Y, Deng Z, Liu X, Liu S, Zhong Y. Src-family kinases activation in spinal microglia contributes to central sensitization and chronic pain after lumbar disc herniation. Mol Pain. 2017 Jan-Dec;13:1744806917733637. doi: 10.1177/1744806917733637. PMID 28952414
- [Background] Akeda K, Takegami N, Yamada J, Fujiwara T, Nishimura A, Sudo A. Central Sensitization in Chronic Low Back Pain: A Population-Based Study of a Japanese Mountain Village. J Pain Res. 2021 May 18;14:1271-1280. doi: 10.2147/JPR.S301924. eCollection 2021. PMID 34040431
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- See also: SF-36 — https://www.physio-pedia.com/36-Item_Short_Form_Survey_(SF-36)